CLINICAL TRIAL: NCT02578277
Title: Effects of BMS-955176 on the Single-dose Pharmacokinetics of Probe Substrates (Caffeine, Metoprolol, Montelukast, Flurbiprofen, Omeprazole, Midazolam, Digoxin, and Pravastatin) in Healthy Subjects
Brief Title: Study on Effects of BMS-955176 on the Pharmacokinetics of Probe Substrates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 206294; AI468-063 (Other: BMS ID)
Record Dates: First submitted 2015-10-15; First posted 2015-10-16 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — BMS-955176

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single sequence, 3-period DDI (drug-drug interaction) (Experimental): Single sequence
  Interventions: Drug: CYP and transporter probe substrates; Drug: BMS-955176; Drug: BMS-955176 plus CYP and transporter probe substrates

INTERVENTIONS:
Drug: CYP and transporter probe substrates — Cocktail of CYP (cytochrome P450) and transporter probe substrates
Drug: BMS-955176 — BMS-955176
Drug: BMS-955176 plus CYP and transporter probe substrates — BMS-955176 plus the cocktail of CYP and transporter probe substrates

SUMMARY:
The purpose of the study is to study the effects of BMS-955176 on the single-dose PK parameters of probe substrates caffeine, metoprolol, montelukast, flurbiprofen, omeprazole, midazolam, digoxin, and pravastatin

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent
2. Healthy male and female (not of childbearing potential) subjects as determined by medical history, surgical history, physical examination, vital signs, ECGs, and clinical laboratory determinations
3. Body mass index (BMI) of 18.0 kg/m2 to 32.0 kg/m2, inclusive, at screening and Day 1. BMI = weight (kg)/[height(m)]
4. Women must have documented proof that they are not of childbearing potential (eg, surgically sterile, postmenopausal with a documented follicle-stimulating hormone (FSH) > 40 mIU/mL) and should not be breast feeding
5. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with BMS-955176 in addition to a post-treatment completion period

Exclusion Criteria:

1. Any significant acute or chronic medical illness
2. Use of tobacco, excessive alcohol
3. Medical history indicative of an increased risk of a cardiac arrhythmia or cardiac disease and history of asthma, bronchospasm, sleep apnea, rhabdomyolysis, a bleeding disorder, a major depressive disorder within the past 6 months, peptic ulcer or significant GI bleed, Raynaud's disease, or any gastrointestinal surgery that could impact upon the absorption of study drug
4. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations beyond what is consistent with the target population
5. History of allergy to BMS-955176, digoxin (or any member of the digitalis glycosides class of drugs), caffeine, metoprolol, montelukast, flurbiprofen, omeprazole, midazolam, or pravastatin, or to any related compounds

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2015-12-23 (Actual); Study Completion 2015-12-23 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum observed concentration) | Days 1 to 18
AUC(0-T), area under the concentration-time curve from time zero to the time of the last quantifiable concentration | Days 1 to 18
AUC(INF), area under the concentration-time curve from time zero extrapolated to infinite time | Days 1 to 18

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States